CLINICAL TRIAL: NCT04805970
Title: REsearching Covid-19 Outcomes in Diabetes (RECODE)
Acronym: RECODE
Status: Active, not recruiting | Type: Observational
Sponsor: AdventHealth Translational Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 1605203
Record Dates: First submitted 2021-03-17; First posted 2021-03-18 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Covid19; Diabetes
MeSH Terms: conditions — COVID-19; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with and without diabetes who were previously diagnosed with COVID-19

SUMMARY:
The purpose of this study is to observe any changes that may occur to certain organs following a confirmed diagnosis of COVID-19 in people with and without diabetes.

ELIGIBILITY:
Inclusion Criteria:

For Type 2 Diabetes (T2D)

1. Male or female 18 years of age and older willing and able to give informed consent to participate in the study
2. Confirmed diagnosis of SARS-CoV-2 RNA via a polymerase chain reaction (PCR) assay (having been discharged at least 2 months from hospital but not greater than 6 months).
3. Diagnosis of T2D according to American Diabetes Association (ADA) criteria.
4. Must have access to a computer/laptop or a modern (no more than 3-4 years old) smart phone/tablet for cognitive assessments.

For participant without Type 2 Diabetes (T2D)

1. Male or female 18 years of age and older willing and able to give informed consent to participate in the study
2. Confirmed diagnosis of SARS-CoV-2 RNA via a polymerase chain reaction (PCR) assay (having been discharged at least 2 months from hospital but not greater than 6 months).
3. Must have access to a computer/laptop or a modern (no more than 3-4 years old) smart phone/tablet for cognitive assessments.

Exclusion Criteria:

1. Symptoms of active respiratory viral infection:

   1. high temperature (over 37.8°C/100.4°F)
   2. cough (consistent for over an hour; 3 or more episodes in 24 hours)
2. Any history of Type I diabetes
3. The participant may not enter the study with any known contraindication to magnetic resonance imaging including

   1. Pregnancy, lactation or 6 months postpartum from the scheduled date of collection
   2. Metal implants (pacemaker, aneurysm clips) based on Investigator's judgment at Screening
   3. Unable to participate in MRI assessments due to physical limitations of equipment tolerances (e.g. MRI bore size) based on Investigator's judgment at Screening
   4. Unable to tolerate MRI imaging or claustrophobia
4. Any condition, including a significant underlying disease or disorder which, in the opinion of the investigator, may put the participant at risk by participating in the study or limit the participant's ability to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who were initially hospitalized with laboratory-confirmed SARS-CoV-2 infection [COVID-19 disease], who are no-longer considered infectious by approved bioassay
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Measure and characterize organ volume change in patients with and without diabetes through use of summary statistics. | 1 year
  Patients recovering from the COVID-19 disease

CONTACTS AND LOCATIONS:
Overall Officials: Richard Pratley, MD, Principal Investigator — AdventHealth Orlando
Locations (1):
- AdventHealth Translational Research Institute, Orlando, Florida, United States